CLINICAL TRIAL: NCT04375826
Title: Continuous Preperitoneal Analgesia Versus Thoracic Epidural Analgesia After Open Pancreaticoduodenectomy: a Randomized Controlled Open-labeled Noninferiority Trial
Brief Title: Preperitoneal Analgesia Versus Epidural Analgesia After Open Pancreaticoduodenectomy
Acronym: Pain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Young Jang, Associate professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2003-128-111
Record Dates: First submitted 2020-04-26; First posted 2020-05-05 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Pain Management; Pain, Postoperative
Keywords: Pain management; Postoperative pain
MeSH Terms: conditions — Agnosia; Pain, Postoperative | interventions — Analgesia, Patient-Controlled

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Epidural analgesia (Active Comparator): Only Epidural analgesia is used for this group
  Interventions: Device: Epidural patient controlled analgesia
- Preperitoneal analgesia and IV-PCA (Active Comparator): This group is given with both preperitoneal analgesia and Intravenous Patient Controlled Analgesia (IV-PCA)
  Interventions: Device: Preperitoneal analgesia and IV-PCA

INTERVENTIONS:
Device: Epidural patient controlled analgesia — The device is connected to the epidural catheter prior to surgery and drug administration is started during surgery. The continuous infusion rate is 4 ml / hr. When the button is pressed, 2 ml is additionally administered and the lock time is 20 minutes.
  Arms: Epidural analgesia
Device: Preperitoneal analgesia and IV-PCA — During surgery, the preperitoneal analgesia catheters are inserted into the preperitoneal space and these catheters are connected to the pump with ropivacaine.
  Arms: Preperitoneal analgesia and IV-PCA

SUMMARY:
This is a prospective randomized open-label noninferiority trial that compares thoracic epidural analgesia and continuous preperitoneal analgesia after open pancreaticoduodenectomy.

DETAILED DESCRIPTION:
In the Enhanced recovery after surgery (ERAS) program of pancreaticoduodenectomy (PD), thoracic epidural analgesia (or epidural analgesia) was considered to be a key analgesic method because it not only effectively controls pain, but also lowers insulin resistance and helps restore bowel movement. However, epidural analgesia can cause a number of side effects despite of effective pain control. Epidural analgesia reduces peripheral vascular resistance by blocking sympathetic nerves with local anesthetics and may cause hypotension and decreasing heart rate. In addition, it can cause orthostatic hypotension, which can interfere with early ambulation after operation. In rare cases, there are potential complications of epidural abscess, meningitis, and epidural hematoma.

Continuous peritoneal analgesia using local anesthetics has recently been used as an alternative analgesic to epidural analgesia in open abdomen surgery. This is easier to perform than epidural analgesia and is known to have fewer side effects. Recently, a non-inferiority comparison study have revealed that peritoneal analgesic was not inferior to epidural analgesia in terms of pain control. However, this study included a variety of operations other than PD, and most of the incisions were substernal, not midline. In addition, the method for mounting the epidural catheter was not described. The failure rate of the epidural catheter was reported to be 15%.

The investigators will examine the effect of continuous peritoneal analgesic postoperative pain control in patients undergoing open PD to improve postoperative pain management and to create an our own ERAS program. To this end, The investigators will test non-inferiority between epidural analgesia and peritoneal analgesia.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Disease of periampullary lesions
* Elective open pancreaticoduodenectomy (PD): PD or pylorus preserving pancreaticoduodenectomy (PPPD)
* Midline incision
* Written informed consent : ability to understand and the willingness to sign a written informed consent
* Performance status (ECOG scale): 0-1 at the time of enrollment
* Physical status (ASA) : 1-2 grade

Exclusion Criteria:

* History of any abdominal surgery (except laparoscopic appendectomy, laparoscopic/robotic cholecystectomy, laparoscopic/robotic obstetrics and gynecology surgeries,Cesarean section, laparoscopic/robotic prostate surgery)
* Emergency operation
* History of chronic pain
* Chronic use of opioid, analgesics, anti-depressant, anti-epileptics (>1year)
* Alcoholics
* Impossible to control PCA d/t delirium, cognitive impairment
* Contraindication for epidural analgesia
* Patients with coagulopathy (INR>1.5, Prothrombin time>1.5, platelets <80x10^9perL) or anti-coagulants
* Hypersensitive to fentanyl and ropivacaine
* Need other organ resection (ex. Liver, colon)
* Intubation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2020-11-13 (Actual); Primary Completion 2023-10-26 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean numerical rating score for pain after operation | 1-3 days after operation
  The scale of the numerical rating score for pain is 0~10 and higher score is worse outcome.
  Mean NRS pain scores are compared between two groups.

SECONDARY OUTCOMES:
Pain related factors | postoperative day 1,2,and 3
  The scale of the numerical rating score for pain is 0~10 and higher score is worse outcome.
  Numerical rating score for pain on postoperative day 1, 2 and 3 at 4pm
QoR-15 Survey | postoperative day 1,2,and 3
  QoR-15 survey on postoperative day 1,2,and 3.
Recovery related factors | Within 1 week after operation
  Time to first eat meal, time to first move, time to first gas out
Postoperative complication factors | Within 1 week after operation
  Clavien-Dindo classification, postoperative pancreatic fistula
analgesic related factors | postoperative day 1,2,and 3
  rescue analgesics amounts, opioid amounts
Opioid related factors | postoperative day 1,2,and 3
  nausea, hypotension, respiratory depression
Hospital stay | at discharge
  postoperative hospital stay day

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Young Jang, M.D., PhD., Study Chair — Seoul National University Hospital
Locations (1):
- Department of Surgery, Seoul National University College of Medicine, Seoul, South Korea

REFERENCES:
- [Derived] Lee M, Jung JY, Han Y, Chae YS, Yun WG, Jung HS, Cho YJ, Choi YJ, Lee HJ, Kwon W, Kim WH, Jang JY. Continuous preperitoneal versus thoracic epidural analgesia in open pancreatoduodenectomy: randomized clinical trial. Br J Surg. 2024 Nov 27;111(12):znae296. doi: 10.1093/bjs/znae296. PMID 39602790